CLINICAL TRIAL: NCT00006170
Title: Bupropion and Weight Control for Smoking Cessation
Brief Title: Bupropion and Weight Control for Smoking Cessation - 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Marsha Marcus, Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-04174-1; R01DA004174 (NIH)
Record Dates: First submitted 2000-08-09; First posted 2000-08-10 (Estimated); Results first posted 2013-11-14 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-06

CONDITIONS: Tobacco Use Disorder
Keywords: smoking cessation; Women; bupropion; weight concerns; weight
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Body Weight | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Bupropion and Weight Concerns intervention (Experimental): Bupropion SR and a weight concerns psychosocial intervention
  Interventions: Drug: Bupropion; Behavioral: weight concerns intervention
- Placebo and Weight Concerns (Active Comparator): A matched placebo administered on same schedule as bupriopion and a weight concerns psychosocial intervention for smoking cesstion
  Interventions: Drug: Placebo; Behavioral: weight concerns intervention
- Bupropion and standard smoking cessation (Active Comparator): Bupropion SR and a time and attention controlled smoking cessation intervention
  Interventions: Drug: Bupropion; Behavioral: smoking cessation intervention
- Placebo and standard smoking cessation (Placebo Comparator): A matched placebo administered on same schedule as bupriopion and a time and attention controlled smoking cessation intervention
  Interventions: Drug: Placebo; Behavioral: smoking cessation intervention

INTERVENTIONS:
Drug: Bupropion — smoking cessation medication aid
  Other Names: zyban
  Arms: Bupropion and Weight Concerns intervention; Bupropion and standard smoking cessation
Drug: Placebo — A matched placebo pill
  Arms: Placebo and Weight Concerns; Placebo and standard smoking cessation
Behavioral: weight concerns intervention — cognitive behavioral treatment to address weight concners
  Arms: Bupropion and Weight Concerns intervention; Placebo and Weight Concerns
Behavioral: smoking cessation intervention — Cognitive behavioral intervention for smoking cessation
  Arms: Bupropion and standard smoking cessation; Placebo and standard smoking cessation

SUMMARY:
The purpose of this study is to determine whether the addition of bupropion (Zyban) to cognitive behavioral therapy (CBT) will enhance longer-term tobacco abstinence in women.

DETAILED DESCRIPTION:
Although rates of smoking have declined, the decrease in prevalence has been much less pronounced in women than in men, and women are particularly vulnerable to ongoing smoking-related morbidity and mortality. One important reason for gender differences in smoking cessation is concern about cessation-related weight gain among women, which is associated with poorer cessation outcome. We previously documented that cognitive behavior therapy to minimize weight concerns (CBT) was effective in promoting cessation and controlling weight gain among weight concerned women smokers. The current study is a randomized, double-blind, controlled trial to determine whether the addition of bupropion (Zyban) to CBT (12 sessions over 14 weeks, with 6 booster sessions) will enhance longer-term abstinence. Bupropion was the clear medication of choice for this trial because it is efficacious in promoting smoking cessation, attenuates cessation-related weight gain (particularly in women), and relieves negative mood, which appears more common in weight-concerned women. Four hundred fifty weight concerned women smokers will be randomized to either CBT for weight concerns plus standard cessation or standard smoking cessation only and six months of either bupropion (Zyban) or placebo (2 x 2 design). Primary outcome will be rates of smoking abstinence at 1 year and time to relapse across the four treatment conditions. In addition, we will determine the effects of these treatments on tobacco withdrawal, mood, and weight. Results of this investigation will provide information on the relative efficacy of the CBT intervention and bupropion alone and in combination and the utility of drug and counseling strategies that are specifically tailored for a high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Smoke at least 10 cigarettes per day
* Report concern about cessation-related weight gain
* Motivated to quit smoking

Exclusion Criteria:

* Currently pregnant, lactating, or no medically approved method of contraception
* Major medical problem
* History of seizure disorder or head injury
* Current or historical psychosis or bipolar disorder
* History of alcohol or substance abuse within previous year
* Current or historical eating disorder
* Use of antidepressant medication, monoamine oxidase inhibitor or lithium with previous month
* Multiple Drug Allergies
* Current major depressive disorder

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2000-09; Primary Completion 2009-12 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marsha Marcus, Ph.D., Principal Investigator — Western Psychiatric Institute & Clinic
Locations (1):
- Western Psychiatric Institute & Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Levine MD, Perkins KA, Kalarchian MA, Cheng Y, Houck PR, Slane JD, Marcus MD. Bupropion and cognitive behavioral therapy for weight-concerned women smokers. Arch Intern Med. 2010 Mar 22;170(6):543-50. doi: 10.1001/archinternmed.2010.33. PMID 20308641
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were recruited between September 1999 and October 2005.
Pre-assignment Details: Potential participants were excluded for current MDD, suicidality, drug or alcohol dependence within the past year, psychotic disorders, conditions associated with lowered seizure threshold, use of medications contraindicated with bupropion, uncontrolled hypertension, recent use of bupropion, pregnancy or use of other smoking or weight treatments.
Groups:
- Weight Concerns + Bupropion (WC+B): An approach was taken to combine cognitive behavioral therapy and pharmacotherapy to women who had weight concerns after cessation. This group took bupropion, a widely used, efficacious smoking cessation agent.
- Weight Concerns + Placebo (WC+P): An approach was taken to combine cognitive behavioral therapy and pharmacotherapy to women who had weight concerns after cessation. This group took a placebo instead of the bupropion.
- Social Support + Bupropion (SS+B): An approach was taken to combine standard cessation therapy with added discussion of smoking topics but no specific weight focus and pharmacotherapy. This group took bupropion, a widely used, efficacious smoking cessation agent.
- Social Support + Placebo (SS+P): An approach was taken to combine standard cessation therapy with added discussion of smoking topics but no specific weight focus and pharmacotherapy. This group took a placebo instead of the bupropion.
Period: Overall Study
Arm/Group | Weight Concerns + Bupropion (WC+B) | Weight Concerns + Placebo (WC+P) | Social Support + Bupropion (SS+B) | Social Support + Placebo (SS+P)
Started | 106 | 87 | 89 | 67
Completed | 57 | 37 | 46 | 28
Not Completed | 49 | 50 | 43 | 39

BASELINE CHARACTERISTICS:
Groups:
- WC+B: An approach was taken to combine cognitive behavioral therapy and pharmacotherapy to women who had weight concerns after cessation. This group took bupropion, a widely used, efficacious smoking cessation agent.
- WC+P: An approach was taken to combine cognitive behavioral therapy and pharmacotherapy to women who had weight concerns after cessation. This group took a placebo instead of bupropion.
- SS+B: An approach was taken to combine standard cessation therapy with added discussion of smoking topics but no specific weight focus and pharmacotherapy. This group took bupropion, a widely used, efficacious smoking cessation agent.
- SS+P: An approach was taken to combine standard cessation therapy with added discussion of smoking topics but no specific weight focus and pharmacotherapy. This group took a placebo instead of the bupropion.
- Total: Total of all reporting groups
Arm/Group | WC+B | WC+P | SS+B | SS+P | Total
Number analyzed (Participants) | 106 | 87 | 89 | 67 | 349
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 106 | 87 | 89 | 67 | 349
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (9.2) | 42.6 (10.0) | 41.0 (11.2) | 42.3 (10.4) | 42.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 87 | 89 | 67 | 349
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 106 | 87 | 89 | 67 | 349

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence
Description: Women were interviewed using the time-line follow-back method and expired-air carbon monoxide (CO) was collected using a Vitalograph BreathCO monitor. Salivary samples were collected immediately after each assessment visit (1, 3, 6, and 12 mo). A CO reading of 8ppm or less and cotinine level of >15 micrograms/L were used to confirm non-smoking.
Time Frame: 3 months
Population: Participants with available data at 3mo. All others were unable to provide data at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | WC+B | WC+P | SS+B | SS+P
Number analyzed (Participants) | 70 | 39 | 56 | 37
percentage of participants | 41 (1) | 18 | 33 | 19
Statistical Analysis 1: Comparison: WC+B vs WC+P; Test type: Non-Inferiority or Equivalence — Power was determined using a log-rank statistic for comparing 2 survival curves, with a 2-sided alpha level of 0.05 and 40% as the reference from which differences were computed; p = 0.001, Regression, Logistic
Statistical Analysis 2: Comparison: WC+B vs SS+B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.25, Regression, Logistic
Statistical Analysis 3: Comparison: SS+B vs SS+P; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.07, Regression, Logistic

2. Primary Outcome: Smoking Abstinence
Description: as for outcome 1
Time Frame: 6 months
Population: Participants with available data at 6mo. All others were unable to provide data at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | WC+B | WC+P | SS+B | SS+P
Number analyzed (Participants) | 64 | 40 | 47 | 32
percentage of participants | 34 | 11 | 21 | 10
Statistical Analysis 1: Comparison: WC+B vs WC+P; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Regression, Logistic
Statistical Analysis 2: Comparison: WC+B vs SS+B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.053, Regression, Logistic
Statistical Analysis 3: Comparison: SS+B vs SS+P; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.08, Regression, Logistic

3. Primary Outcome: Smoking Abstinence
Description: as for outcome 1
Time Frame: 12 months
Population: Participants with available data at 12mo. All others were unable to provide data at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | WC+B | WC+P | SS+B | SS+P
Number analyzed (Participants) | 57 | 37 | 46 | 28
percentage of participants | 24 | 8 | 19 | 7
Statistical Analysis 1: Comparison: WC+B vs WC+P; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.006, Regression, Logistic
Statistical Analysis 2: Comparison: WC+B vs SS+B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.45, Regression, Logistic
Statistical Analysis 3: Comparison: SS+B vs SS+P; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.046, Regression, Logistic

ADVERSE EVENTS:
Arm/Group | WC+B | WC+P | SS+B | SS+P
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/87 | 0/89 | 0/67
Other Adverse Events (participants affected / at risk) | 0/106 | 0/87 | 0/89 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No